CLINICAL TRIAL: NCT05704595
Title: Effectiveness of Outpatient Intravenous Diuretic Therapy for Treatment of Worsening Heart Failure (OUTPATIENT-WHF)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study no longer moving forward
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00111091
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial outpatient management strategy, including outpatient IV diuretics in clinic (Other)
  Interventions: Other: Initial outpatient management strategy, including outpatient IV diuretics in clinic
- Initial hospitalization-based management strategy (Other)
  Interventions: Other: Initial hospitalization-based management strategy

INTERVENTIONS:
Other: Initial outpatient management strategy, including outpatient IV diuretics in clinic — Management strategy including IV diuretic in the outpatient clinic
  Arms: Initial outpatient management strategy, including outpatient IV diuretics in clinic
Other: Initial hospitalization-based management strategy — Direct admission to the hospital
  Arms: Initial hospitalization-based management strategy

SUMMARY:
The purpose of the OUTPATIENT-WHF study is to characterize the effectiveness of outpatient intravenous diuretic therapy as a treatment for worsening heart failure.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether treating certain patients with worsening heart failure as an outpatient with intravenous and oral medications can work just as well as treating patients in the hospital.

Participants who enter into the study and meet eligibility criteria will be randomly chosen to either get intravenous diuretic like Lasix in the clinic and get outpatient care, versus directly admitted to the hospital to receive intravenous diuretic and normal hospital care.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Presentation to a Duke outpatient clinic with heart failure requiring IV diuretics, as per clinician judgement
3. Able to provide signed informed consent
4. Successful completion of EuroQOL-5 dimensions survey

Exclusion Criteria:

1. Managing clinician without equipoise for initial outpatient treatment strategy versus initial hospitalization-based treatment strategy for heart failure, and decline to accept randomization.
2. Patient without equipoise for initial outpatient treatment strategy versus initial hospitalization-based treatment strategy for heart failure, and decline to accept randomization.
3. History of left ventricular assist device or heart transplantation
4. End-stage kidney disease requiring chronic dialysis therapy
5. New diagnosis of heart failure
6. Pregnant or breast-feeding
7. Fever >101.0 degrees Fahrenheit at screening
8. Any other condition that in the judgment of the investigator would jeopardize the patient's compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital | 30 days

SECONDARY OUTCOMES:
Days alive and out of hospital | 90 days
Total hospitalizations | 30 days
Total hospitalizations | 90 days
Total emergency department visits | 30 days
Total emergency department visits | 90 days
Death | 30 days
Death | 90 days
Health status as measured by EuroQOL-5 dimensions (EQ5D) utility index | 30 days
  The EQ5D utility index consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories (no problems, slight problems, moderate problems, severe problems, and extreme problems), from which a single EQ-5D index score can be calculated ranging from 0 (dead) to 1 (perfect health).
Health status as measured by EuroQOL-5 dimensions (EQ5D) visual analog scale (VAS) | 30 days
  The EQ5D VAS measures one's self-perceived health today on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health) on which participants have to indicate their current health.
Health status as measured by EuroQOL-5 dimensions (EQ5D) utility index | 90 days
  The EQ5D utility index consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories (no problems, slight problems, moderate problems, severe problems, and extreme problems), from which a single EQ-5D index score can be calculated ranging from 0 (dead) to 1 (perfect health).
Health status as measured by EuroQOL-5 dimensions (EQ5D) visual analog scale (VAS) | 90 days
  The EQ5D VAS measures one's self-perceived health today on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health) on which participants have to indicate their current health.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Greene, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No